CLINICAL TRIAL: NCT05687474
Title: Universal Genomic Newborn Screening in the Wallonia-Brussels Federation: Baby Detect
Brief Title: Baby Detect : Genomic Newborn Screening
Acronym: BabyDetect
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other); University of Liege (Other); Sanofi (Industry); Orchard Therapeutics (Industry); Takeda (Industry); Zentech-Lacar Company (Unknown); Leon Fredericq Foundation (Unknown)
Responsible Party: Principal Investigator, Laurent Servais, Professor, Centre Hospitalier Universitaire de Liege
Other Study IDs: Baby Detect
Record Dates: First submitted 2022-12-28; First posted 2023-01-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Congenital Adrenal Hyperplasia; Familial Hyperinsulinemic Hypoglycemia 1; Phosphoglucomutase 1 Deficiency; Maturity Onset Diabetes of the Young; Cystic Fibrosis; Hypophosphatasia, Infantile; Congenital Hypothyroidism; Deficit in Anterior Pituitary Function and Variable Immunodeficiency; Pituitary Hormone Deficiency, Combined; Diamond Blackfan Anemia; Wiskott-Aldrich Syndrome; Fanconi Anemia; Hemophilia A; Hemophilia B; Glucose 6 Phosphate Dehydrogenase Deficiency; Alpha-Thalassemia; Sickle Cell Disease; Shwachman-Diamond Syndrome; Alpha 1-Antitrypsin Deficiency; Inflammatory Bowel Disease 25, Autosomal Recessive; Wilson Disease; Progressive Familial Intrahepatic Cholestasis; Crigler-Najjar Syndrome; Familial Chylomicronemia; Lysosomal Acid Lipase Deficiency; Familial Hemophagocytic Lymphocytosis; Griscelli Syndrome; Chediak-Higashi Syndrome; Severe Congenital Neutropenia; Severe Combined Immune Deficiency; Chronic Granulomatous Disease; Menkes Disease; Adrenoleukodystrophy; Smith-Lemli-Opitz Syndrome; Ataxia With Vitamin E Deficiency; Thiamine Metabolism Dysfunction Syndrome 5 (Episodic Encephalopathy Type); Thiamine Metabolism Dysfunction Syndrome 4 (Bilateral Striatal Degeneration and Progressive Polyneuropathy Type); Thiamine-Responsive Megaloblastic Anemia; Thiamine Metabolism Dysfunction Syndrome 2; Deficiency of GOT2; Cerebral Folate Transport Deficiency; Segawa Syndrome, Autosomal Recessive; Congenital Myasthenic Syndrome; Metachromatic Leukodystrophy; Sepiapterin Reductase Deficiency; Dopamine Beta Hydroxylase Deficiency; Glut1 Deficiency Syndrome; Late-Infantile Neuronal Ceroid Lipofuscinosis; Aromatic L-amino Acid Decarboxylase Deficiency; Charcot-Marie-Tooth Disease, Type 6C; Hereditary Hyperekplexia; Brain Dopamine-Serotonin Vesicular Transport Disease; Very Long Chain Hydroxy Acyl Dehydrogenase Deficiency; Tyrosinemia, Type I; Disaccharide Intolerance I; Beta Ketothiolase Deficiency; Phosphoglycerate Dehydrogenase Deficiency; Succinyl-Coa:3-Ketoacid Coa-Transferase Deficiency; Pyridoxine-5'-Phosphate Oxidase Deficiency; Pyridoxine-Dependent Epilepsy; Propionic Acidemia; Pompe Disease; Phenylalanine Hydroxylase Deficiency; Ornithine Transcarbamylase Deficiency; N Acetyl Glutamate Synthetase Deficiency; Riboflavin Deficiency; Maple Syrup Urine Disease; Medium Chain Acyl CoA Dehydrogenase Deficiency; Malonic Acidemia; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; Isovaleric Acidemia; Phosphoserine Aminotransferase Deficiency; Phosphoserine Phosphatase Deficiency; Hyperornithinemia-Hyperammonemia-Homocitrullinuria; S-Adenosylhomocysteine Hydrolase Deficiency; Mucopolysaccharidosis VII; Mucopolysaccharidosis VI; Mucopolysaccharidosis IV A; Mucopolysaccharidosis II; Mucopolysaccharidosis I; Transcobalamin Deficiency; Isolated Methylmalonic Acidemia; Cobalamin Deficiency; Homocystinuria; Holocarboxylase Synthetase Deficiency; Fanconi Bickel Syndrome; Glycogen Storage Disease; Glycine Encephalopathy; Glutaric Acidemia I; Glucose Galactose Malabsorption; Gaucher Disease, Type 1; Galactosemias; Fructosemia; Fructose-1,6-Diphosphatase Deficiency; Carbamoyl Phosphate Synthase 1 Deficiency; Citrullinemia Type II; Citrullinemia 1; Creatine Deficiency Syndrome; Systemic Primary Carnitine Deficiency; Carnitine Palmitoyltransferase Deficiency 2; Carnitine Palmitoyltransferase Deficiency 1; Carnitine Acylcarnitine Translocase Deficiency; Riboflavin Transporter Deficiency; Branched-Chain Keto Acid Dehydrogenase Kinase Deficiency; Andersen Tawil Syndrome; Timothy Syndrome; Jervell-Lange Nielsen Syndrome; Catecholaminergic Polymorphic Ventricular Tachycardia; Familial Hypertrophic Cardiomyopathy Type 4; Pseudohypoaldosteronism, Type II; Pseudohypoaldosteronism Type 1; Primary Hyperoxaluria; X Linked Hypophosphatemia; Hereditary Nephrogenic Diabetes Insipidus; Cystinosis; Congenital Nephrotic Syndrome, Finnish Type; Alport Syndrome; Hereditary Retinoblastoma; Biotinidase Deficiency; Aciduria, Argininosuccinic; Argininemia; Acyl-CoA Dehydrogenase Family, Member 9, Deficiency of; 3-Hydroxy 3-Methyl Glutaric Aciduria; 3-Hydroxy-3-Methylglutaryl-CoA Synthase 2 Deficiency
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Congenital Hyperinsulinism; Glycogen Storage Disease XIV; Diabetes Mellitus, Type 2; Cystic Fibrosis; Hypophosphatasia, Infantile; Congenital Hypothyroidism; Combined Pituitary Hormone Deficiency; Anemia, Diamond-Blackfan; Wiskott-Aldrich Syndrome; Fanconi Anemia; Hemophilia A; Hemophilia B; Glucosephosphate Dehydrogenase Deficiency; alpha-Thalassemia; Anemia, Sickle Cell; Shwachman-Diamond Syndrome; alpha 1-Antitrypsin Deficiency; Inflammatory Bowel Disease 25, Autosomal Recessive; Hepatolenticular Degeneration; Cholestasis, progressive familial intrahepatic 1; Crigler-Najjar Syndrome; Hyperlipoproteinemia Type I; Wolman Disease; Lymphohistiocytosis, Hemophagocytic; Chediak-Higashi Syndrome; Neutropenia, Severe Congenital, Autosomal Recessive 3; Severe Combined Immunodeficiency; Granulomatous Disease, Chronic; Menkes Kinky Hair Syndrome; Adrenoleukodystrophy; Smith-Lemli-Opitz Syndrome; Ataxia with vitamin E deficiency; Basal ganglia disease, biotin-responsive; Neurodegeneration Due To Cerebral Folate Transport Deficiency; Segawa syndrome, autosomal recessive; Myasthenic Syndromes, Congenital; Leukodystrophy, Metachromatic; Dystonia, Dopa-Responsive, due to Sepiapterin Reductase Deficiency; dopamine beta hydroxylase deficiency; Glut1 Deficiency Syndrome; Neuronal Ceroid-Lipofuscinoses; Aromatic amino acid decarboxylase deficiency; Charcot-Marie-Tooth Disease; Stiff-Person Syndrome; Tyrosinemias; Sucrase-isomaltase deficiency, congenital; Beta ketothiolase deficiency; Phosphoglycerate Dehydrogenase Deficiency; Succinyl-CoA:3-oxoacid CoA transferase deficiency; Pyridoxamine 5-Prime-Phosphate Oxidase Deficiency; Pyridoxine-dependent epilepsy; Propionic Acidemia; Glycogen Storage Disease Type II; Phenylketonurias; Ornithine Carbamoyltransferase Deficiency Disease; Aspartylglucosaminuria; Riboflavin Deficiency; Maple Syrup Urine Disease; Medium chain acyl CoA dehydrogenase deficiency; Malonic aciduria; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Acidemia, isovaleric; Phosphoserine Aminotransferase Deficiency; HHH syndrome; Hypermethioninemia; Mucopolysaccharidosis VII; Mucopolysaccharidosis VI; Mucopolysaccharidosis IV; Mucopolysaccharidosis II; Mucopolysaccharidosis I; Methylmalonic acidemia; Vitamin B 12 Deficiency; Homocystinuria; Holocarboxylase Synthetase Deficiency; Fanconi Syndrome; Glycogen Storage Disease; Hyperglycinemia, Nonketotic; Glutaric Acidemia I; Glucose-Galactose Malabsorption; Gaucher Disease; Galactosemias; Fructose Intolerance; Fructose-1,6-Diphosphatase Deficiency; Carbamoyl-Phosphate Synthase I Deficiency Disease; Neonatal-onset citrullinemia type 2; Citrullinemia; Systemic carnitine deficiency; Carnitine palmitoyl transferase 2 deficiency; Carnitine palmitoyl transferase 1A deficiency; Carnitine-Acylcarnitine Translocase Deficiency; Brown-Vialetto-Van Laere syndrome; Andersen Syndrome; Timothy syndrome; Jervell-Lange Nielsen Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Cardiomyopathy, Familial Hypertrophic, 4; Pseudohypoaldosteronism; Hyperoxaluria, Primary; Familial Hypophosphatemic Rickets; Diabetes Insipidus, Nephrogenic; Cystinosis; Nephrosis, congenital; Nephritis, Hereditary; Retinoblastoma; Biotinidase Deficiency; Argininosuccinic Aciduria; Hyperargininemia; Acyl-CoA Dehydrogenase Family, Member 9, Deficiency of; 3-Hydroxy-3-Methylglutaryl-CoA Lyase Deficiency; 3-Hydroxy-3-Methylglutaryl-CoA Synthase 2 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 drops of dried blood on a blotter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newborns with consent: Newborns with parent's consent

SUMMARY:
Newborn screening (NBS) is a global initiative of systematic testing at birth to identify babies with pre-defined severe but treatable conditions. With a simple blood test, rare genetic conditions can be easily detected, and the early start of transformative treatment will help avoid severe disabilities and increase the quality of life.

Baby Detect Project is an innovative NBS program using a panel of target sequencing that aims to identify 126 treatable severe early onset genetic diseases at birth caused by 361 genes. The list of diseases has been established in close collaboration with the Paediatricians of the University Hospital in Liege. The investigators use dedicated dried blood spots collected between the first day and 28 days of life of babies, after a consent sign by parents.

DETAILED DESCRIPTION:
Every year, thousands of children around the world are born with rare genetic diseases leading to death or lifelong disability. With technological advancements in the field of genetics and medicine, the rate of introduction of treatments for these rare conditions has grown remarkably.

However, timing is of great importance for medication administration. The benefit that can be measured in a patient who has already suffered from a long irreversible degenerative disorder is small and, sometimes, it hardly justifies the cost and the burden of the treatment. Early diagnosis is, thus, of primary importance both to obtain the best effect of the innovative medications and to accelerate their development.

The investigators are pioneered in the field of genetic newborn screening (NBS) in rare diseases by funding, designing, and leading an innovative genetic NBS program initiated in March 2018 in Southern Belgium for Spinal Muscular Atrophy (SMA) that allowed, so far, for 11 children to be detected and treated early and avoid the terrible fate of the disease. The program was disseminated in 17 countries and included public dissemination and health-economic analysis since the very beginning [1]. (www.facebook.com/sunmayariseonsma).

Drawing upon our experience with SMA screening, the investigators have designed a project to screen up to 40,000 newborns/year progressively in 3 years for virtually all the rare diseases that can benefit from treatment or a pre-symptomatic clinical trial.

The methodology of Baby Detect includes sequencing of target genes on dried blood spots collected from the NBS cards in a timely and cost-efficient manner, and its high dynamicity allows for any newly treatable rare disease to be included in its scheme in no longer than 6 months.

Baby Detect, as a multidisciplinary newborn screening program, involves expertise in areas from genetics and medicine to laboratory studies, computer science, Data Protection, Ethics, and health economy. It will constitute the proof of concept that is needed before moving to a whole region-scale population.

ELIGIBILITY:
Inclusion Criteria:

* newborn between birth and 28 days of life
* consent of parent

Exclusion Criteria:

* + 28 days
* Non consent of parent

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns whose mothers and/or the second-parents meet the inclusion criteria and have provided their consent to take part in the study
Sampling Method: Non-Probability Sample
Enrollment: 6824 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Acceptability | through study completion, an average of 1 year
  The percentage of parents accepting the proposed screening in comparison with the number of mothers approached for consent
Feasibility - timing | through study completion, an average of 1 year
  The Turn-around time for the different mutations that are screened
Feasibility - reliability | through study completion, an average of 1 year
  The percentage of false positives and the predicted value for each test The estimation of the false negatives through collaboration with physicians treating the different diseases.

SECONDARY OUTCOMES:
Consequence of NBS on early treatment access - timing | through study completion, an average of 1 year
  The time passed between the birth of diagnostic-positive newborns to the initiation of their treatment
Consequence of NBS on early treatment access - frequency | through study completion, an average of 1 year
  The number of patients offered early treatment
To improve the detection technique for disease related mutations that are not detected in classical screening by improving the classification of unspecified variants. | through study completion, an average of 1 year
  The number of new mutations implemented yearly in the NBS.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CRMN, Hôpital La Citadelle, Liège, Wallonia, Belgium

REFERENCES:
- [Background] Boemer F, Hovhannesyan K, Piazzon F, Minner F, Mni M, Jacquemin V, Mashhadizadeh D, Benmhammed N, Bours V, Jacquinet A, Harvengt J, Bulk S, Dideberg V, Helou L, Palmeira L, Dangouloff T; BabyDetect Expert Panel; Servais L. Population-based, first-tier genomic newborn screening in the maternity ward. Nat Med. 2025 Apr;31(4):1339-1350. doi: 10.1038/s41591-024-03465-x. Epub 2025 Jan 28. PMID 39875687
- [Background] Dangouloff T, Hovhannesyan K, Mashhadizadeh D, Minner F, Mni M, Helou L, Piazzon F, Palmeira L, Boemer F, Servais L. Feasibility and Acceptability of a Newborn Screening Program Using Targeted Next-Generation Sequencing in One Maternity Hospital in Southern Belgium. Children (Basel). 2024 Jul 30;11(8):926. doi: 10.3390/children11080926. PMID 39201861
- See also: Related Info — http://www.babydetect.com